CLINICAL TRIAL: NCT02847013
Title: The Use of Liposomal Bupivacaine in TAP Blocks for Women Undergoing Cesarean Section
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jaimey M. Pauli, MD, OB/GYN Resident, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00005133
Record Dates: First submitted 2016-07-25; First posted 2016-07-27 (Estimated); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Pain
Keywords: Postcesarean Section; Postoperative
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo- Tap block w normal saline (Placebo Comparator): After completion of surgery with closer of skin incision a TAP block will be performed. On confirmation of entering the fascial plane, 20cc of Normal saline will be injected after negative aspiration. That will complete the intervention. 20 patients will be in this arm
  Interventions: Procedure: TAP block w normal saline
- Intervention-Tap block w Liposomal bupivacaine (Experimental): After completion of surgery w closure of skin incision a TAP block will be performed. On confirmation of entering the fascial plane, Liposomal bupivacaine 0.33% (10 ml diluted to 20 ml using sterile normal saline) will be injected after negative aspiration. That will complete the intervention. 20 patients will be in this arm
  Interventions: Drug: TAP block w Liposomal bupivacaine

INTERVENTIONS:
Drug: TAP block w Liposomal bupivacaine — TAP block w Liposomal bupivacaine diluted to 0.66% (20 mLs)
  Other Names: Exparel
  Arms: Intervention-Tap block w Liposomal bupivacaine
Procedure: TAP block w normal saline — TAP block w normal saline -preservative free 0.9% sodium chloride (20mLs)
  Arms: Placebo- Tap block w normal saline

SUMMARY:
This present investigation aims to determine whether a transversus abdominous plane(TAP) block, utilizing liposomal bupivacaine (Exparel), at the conclusion of a cesarean section decreases post-operative pain. The hypothesis is that performance of the TAP block with liposomal bupivacaine will decrease post-operative narcotic use.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years of age
* Scheduled cesarean section with or without bilateral tubal ligation
* Planned performance of a Pfannenstiel incision
* Patients are schedule to have a cesarean section with a member of the Women's Health or Maternal and Fetal Medicine Departments at Penn State University Hershey S. Medical Center

Exclusion Criteria:

* History of opioid use
* History of chronic pain syndrome
* Use of general anesthesia during cesarean delivery
* Postoperative SICU admission
* Postpartum hemorrhage (defined as an Estimated Blood Loss of greater then 1,000mL upon completion of the cesarean section)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2019-12-17 (Actual)

PRIMARY OUTCOMES:
Postoperative narcotic use | initial 48 hours postoperatively
  Patient use of standard postoperative narcotics (percocet) will be measured.

SECONDARY OUTCOMES:
Subjective pain scores using 1-10 VAS system | initial 48 hours postoperatively
  Subjective pain scores using 1-10 VAS system will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Jaimey Pauli, MD, Principal Investigator — Milton S. Hershey Medical Center
Locations (1):
- Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided